CLINICAL TRIAL: NCT05417659
Title: The Effect of Suppression of Adipose Lipolysis on GLP-1 and Energy Intake in Men and Women
Brief Title: Glycogen and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Louise Bradshaw, PhD Student, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EIRA1-7142
Record Dates: First submitted 2022-05-17; First posted 2022-06-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2023-10

CONDITIONS: Energy Intake
MeSH Terms: interventions — Exercise; Carbohydrates; Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): A placebo drink to be consumed 1 hour prior to exercise and every 15 minutes during exercise and placebo tablets to be consumed 30 minutes prior to exercise, at the onset of exercise and 30 minutes into exercise.
  Interventions: Other: Placebo
- Exercise plus carbohydrate (Active Comparator): A high carbohydrate drink (1.6g/kg) to be consumed 1 hour prior to exercise and further drinks (0.2g/kg) every 15 minutes during exercise.
  Interventions: Dietary Supplement: Exercise plus carbohydrate
- Exercise plus niacin (Experimental): A dose of niacin (10mg/kg) to be consumed 30 minutes prior to exercise and two further doses (5mg/kg) at the onset of exercise and 30 minutes into exercise.
  Interventions: Dietary Supplement: Exercise plus niacin

INTERVENTIONS:
Dietary Supplement: Exercise plus carbohydrate — A high carbohydrate drink to be consumed 1 hour prior to exercise and every 15 minutes during exercise.
  Arms: Exercise plus carbohydrate
Dietary Supplement: Exercise plus niacin — A dose of niacin to be consumed 30 minutes prior to exercise, at onset of exercise and 30 minutes into exercise.
  Arms: Exercise plus niacin
Other: Placebo — A placebo drink to be consumed 1 hour prior to exercise and every 15 minutes during exercise and placebo tablets to be consumed 30 minutes prior to exercise, at the onset of exercise and 30 minutes into exercise.
  Arms: Control

SUMMARY:
Obesity is the outcome of chronic excessive energy intake and reduced energy expenditure leading to energy imbalance. It is a risk factor for many preventable diseases such as metabolic disease and its consequences such as type 2 diabetes and cardiovascular disease. Sedentary adults have been shown to have an increased appetite in excess of energy requirements and adults who are more active are able to better regulate energy intake. It is thought that carbohydrate availability and specifically hepatic glycogen utilisation during exercise is a regulator of appetite. However, the majority of research so far does not support this theory, potentially due to research not examining the tissue-specific link between glycogen use and appetite. The aim of this study is to assess whether altering substrate utilisation during exercise by suppressing lipolysis influences GLP-1 levels and caloric intake post exercise. Additionally, the study will explore if there is a tissue specific link between substrate utilisation and post exercise energy intake and examine potential sex differences.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-60 and premenopausal women
* Physically active (at least 30 minutes of exercise 3 times a week)
* Body mass index 18.0-30.0 kg·m-2

Exclusion Criteria:

* Weight instability (>5kg change in body mass over last 6 months)
* Restrained eater (e.g. limiting food intake, calorie counting)
* Current smoker
* Aversion or allergy to test meal foods
* Pregnant or lactating
* Amenorrhoea in women
* Any medical condition or medication that could introduce bias into the study (e.g., diabetes, CVD, lipid or glucose metabolism altering medications)
* Any cardiopulmonary condition prohibiting exercise testing
* Any contraindication to niacin or aspirin (e.g., diabetes, gout, clotting disorders, allergy to non-steroidal anti-inflammatory drugs)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Difference in ad libitum energy intake | 2 hours post exercise
  Difference between ad libitum energy intake (kcal) post exercise between trials

OTHER OUTCOMES:
Change in plasma GLP-1 concentrations post exercise | 2 hours
  Incremental area under the curve of plasma GLP-1 concentrations
Change in plasma leptin concentrations post exercise | 2 hours
  Incremental area under the curve of plasma leptin concentrations
Change in plasma insulin concentrations during exercise | 1 hour
  Incremental area under the curve for plasma insulin concentrations
Change in plasma non-esterified fatty acid concentrations during exercise | 1 hour
  Incremental area under the curve for plasma non-esterified fatty acid concentrations
Change in plasma glucose concentrations during exercise | 1 hour
  Incremental area under the curve for plasma glucose concentrations
Change in plasma lactate concentrations during exercise | 1 hour
  Incremental area under the curve for plasma lactate concentrations
Change in carbohydrate oxidation during exercise | 1 hour
  Incremental area under the curve for carbohydrate oxidation
Change in fat oxidation during exercise | 1 hour
  Incremental area under the curve for fat oxidation
Change in skin temperature during exercise | 1 hour
  Incremental area under the curve for skin temperature
Change in core body temperature during exercise | 1 hour
  Incremental area under the curve for core body temperature
Muscle glycogen utilisation | 1 hour
  Difference in muscle glycogen utilisation during exercise between conditions
Extra-muscular glycogen oxidation | 1 hour
  Difference in extra muscular glycogen oxidation during exercise between conditions
Difference in blood pressure between conditions | 3 hours
  Difference in blood pressure between conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided